CLINICAL TRIAL: NCT03754192
Title: Prediction Value of Perfusion and Dual Energy Computer Tomography for Microvascular Invasion in Hepatocellular Carcinoma
Brief Title: Perfusion and Dual Energy Computer Tomography in Hepatocellular Carcinoma
Acronym: PERCAHEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP180011
Record Dates: First submitted 2018-11-14; First posted 2018-11-27 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Perfusion computer tomography; dual-energy computer tomography
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Cytidine Triphosphate

STUDY DESIGN:
Intervention Model Description: Dual-energy computed tomography and perfusion computed tomography
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- perfusion computed tomography (Other): Will be realsed before liver surgery
  Interventions: Radiation: perfusion Computed Tomography

INTERVENTIONS:
Radiation: perfusion Computed Tomography — Will be carried before liver surgery
  Other Names: Computed tomography

SUMMARY:
The aim of this study is to evaluate the hepatic perfusion computer tomography and dual energy computer tomography in the assessment of tumor characterization of Hepatocellular carcinoma in patients with resectable Hepatocellular carcinoma by comparing the quantitative parameters computer tomography obtained with the pathological data of the surgical specimens.

DETAILED DESCRIPTION:
Dual-energy computer tomography and perfusion computer tomography (General Electric revolution Hight definition Gemstone™ Spectral Imaging) will be performed in all patients. Iodine concentration and quantitative perfusion parameters of the Hepatocellular carcinoma and surrounding liver parenchyma data will be compared with the pathological results.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Hepatocellular carcinoma made according to the guidelines of the American Association for the study of the Liver
* Affiliation to a national health insurance
* An indication for hepatic resection during the decision-making stage
* A request for a pre-operative Computer Tomography in our radiology unit
* An affiliation to a social security
* Informed consent given by the patient

Exclusion Criteria:

* Previous treatments of Hepatocellular carcinoma (medicated or surgical)
* Patient under tutorship or curatorship
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Pefusion parameters | 5 minutes
  correlation between pre-operative imaging data and histological data of Hepatocellular carcinoma

SECONDARY OUTCOMES:
Pathological examination | 1 month
  Compare data obtained in perfusion computer tomography to the imaging data and to the Histological differentiation grades

CONTACTS AND LOCATIONS:
Overall Officials: LEWIN MAITE, MD, PhD, Principal Investigator — APHP
Locations (1):
- CHU Paul Brousse, Villejuif, France

REFERENCES:
- [Derived] Lewin M, Laurent-Bellue A, Desterke C, Radu A, Feghali JA, Farah J, Agostini H, Nault JC, Vibert E, Guettier C. Evaluation of perfusion CT and dual-energy CT for predicting microvascular invasion of hepatocellular carcinoma. Abdom Radiol (NY). 2022 Jun;47(6):2115-2127. doi: 10.1007/s00261-022-03511-7. Epub 2022 Apr 13. PMID 35419748